CLINICAL TRIAL: NCT03214705
Title: Role of Computed Tomography Perfusion in Detection of Patients at Risk for Delayed Cerebral Ischemia After Subarachnoid Hemorrhage
Brief Title: Role of CT Perfusion in Predicting Poor Outcome After Subarachnoid Hemorrhage
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel-Tawab Mohamed, Assistant Lecturer, Assiut University
Other Study IDs: CTP predicts DCI
Record Dates: First submitted 2017-06-29; First posted 2017-07-11 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm; Delayed Cerebral Ischemia
Keywords: CT perfusion; Subarachnoid hemorrhage; Vasospasm; Delayed cerebral ischemia
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with poor outcome: Follow up of patients is done for 21 days by combined clinical and radiological examination. Poor clinical outcome is associated with vasospasm leading to permanent neurological deficit, stroke or death.
- Patients without poor outcome: Patients who do not develop delayed cerebral ischemia or stroke, confirmed by combined clinical and radiological examination.

SUMMARY:
Prospective evaluation of patients with subarachnoid hemorrhage (SAH) will be done by computed tomography angiography (CTA) and perfusion imaging (CTP) for any correlation between degree of vasospasm and perfusion deficit as well as evaluating the ability of CTP to predict delayed cerebral ischemia.

DETAILED DESCRIPTION:
Cerebral vasospasm is a serious complication of subarachnoid haemorrhage . In the first 2 weeks of SAH, angiographic vasospasm is seen up to 40-70% of patients and causes ischemic deficits in 15-36% of patients.

The best clinical indicator of significantly reduced brain perfusion (cerebral blood flow (CBF)<20 ml per 100 g/min) is the presence of new neurologic deficits. However, clinical symptoms may be vague and mimic other conditions in patients with SAH.

CT Perfusion can be used in the evaluation of patients with possible vasospasm after subarachnoid hemorrhage (SAH). It can thus be used to assess cerebral ischemia and infarction as a result of vasospasm after SAH.

The presence of cerebral vasospasm identified with transcranial Doppler, digital subtraction angiography, or CT angiography (CTA) is frequently used to confirm DCI. Presence of vasospasm, however, does not prove the presence of ischemia and absence of vasospasm does not rule out. Better diagnostic tests in the acute stage of deterioration, possibly caused by DCI, are therefore needed. In patients with SAH, CTP has recently been shown to be promising for detection of early ischemia.

ELIGIBILITY:
Inclusion Criteria:

* All patients presented with subarachnoid haemorrhage

Exclusion Criteria:

* Patients with abnormal renal functions with creatinine ≥ 2 mg/dl/
* Patients with hypersensitivity to contrast media.
* Contraindication to radiation as pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having subarachnoid hemorrhage whether post aneurysmal or spontaneous
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow (CBF) on Admission | 3 days from the attack
  Cerebral blood flow (CBF) on Admission in units of ml/100 gram brain tissue/ minute.
  The measurements will be compared with the outcome of the patient (namely monitoring delayed cerebral ischemia in SAH patients) to test if early CT perfusion could predict the poor outcome in SAH patients.
Cerebral blood volume (CBV) on Admission | 3 days from the attack
  Cerebral blood volume (CBF) on Admission in units of ml/100 gram brain tissue.
Mean transit time (MTT) on Admission | 3 days from the attack
  Mean transit time (MTT) on Admission in units of seconds.

SECONDARY OUTCOMES:
Correlation of vasospasm to perfusion abnormality using Comparing between CT angiography and CT perfusion in patients with subarachnoid hemorrhage | 4-14 days from the attack
  Evaluating results of CT angiography and CT perfusion in patients for Correlating vasospasm and perfusion abnormality. Results will be dichotomous; positive and negative, then tested by cross tabulation.
Hunt and Hess scale | 3 days from the attack
  Hunt and Hess clinical scale was performed for every patient.
  Grades are as the following:
  Grade 1: Asymptomatic or mild headache Grade 2: Cranial nerve palsy or moderate to severe headache/nuchal rigidity Grade 3: Mild focal deficit, lethargy, or confusion Grade 4: Stupor and/or hemiparesis Grade 5: Deep coma, decerebrate posturing, moribund appearance
Fisher scale | 3 days from the attack
  Fisher scale quantifies the amount of SAH as the following:
  1. None evident
  2. Less than 1 mm thick
  3. More than 1 mm thick
  4. Diffuse or none with intraventricular hemorrhage or parenchymal extension

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel-Tawab, Principal Investigator — Assiut University; Afaf A. Hasan, Profosser, Study Chair — Assiut University; Mohamed A. Ahmed, Professor, Study Director — Assiut University; Hany M. Seif, Professor, Study Director — Assiut University; Hazem A. Youssef, Professor, Study Director — Assiut unviersity
Locations (1):
- Mohamed Abdel-Tawab Mohamed, Asyut, Egypt

REFERENCES:
- [Background] Aralasmak A, Akyuz M, Ozkaynak C, Sindel T, Tuncer R. CT angiography and perfusion imaging in patients with subarachnoid hemorrhage: correlation of vasospasm to perfusion abnormality. Neuroradiology. 2009 Feb;51(2):85-93. doi: 10.1007/s00234-008-0466-7. Epub 2008 Oct 11. PMID 18850093
- [Background] Binaghi S, Colleoni ML, Maeder P, Uske A, Regli L, Dehdashti AR, Schnyder P, Meuli R. CT angiography and perfusion CT in cerebral vasospasm after subarachnoid hemorrhage. AJNR Am J Neuroradiol. 2007 Apr;28(4):750-8. PMID 17416833
- [Background] Dankbaar JW, de Rooij NK, Rijsdijk M, Velthuis BK, Frijns CJ, Rinkel GJ, van der Schaaf IC. Diagnostic threshold values of cerebral perfusion measured with computed tomography for delayed cerebral ischemia after aneurysmal subarachnoid hemorrhage. Stroke. 2010 Sep;41(9):1927-32. doi: 10.1161/STROKEAHA.109.574392. Epub 2010 Aug 5. PMID 20689085
- [Background] Munoz-Guillen NM, Leon-Lopez R, Tunez-Finana I, Cano-Sanchez A. From vasospasm to early brain injury: new frontiers in subarachnoid haemorrhage research. Neurologia. 2013 Jun;28(5):309-16. doi: 10.1016/j.nrl.2011.10.015. Epub 2012 Jan 21. English, Spanish. PMID 22264777
- [Background] Wintermark M, Sincic R, Sridhar D, Chien JD. Cerebral perfusion CT: technique and clinical applications. J Neuroradiol. 2008 Dec;35(5):253-60. doi: 10.1016/j.neurad.2008.03.005. Epub 2008 May 7. PMID 18466974